CLINICAL TRIAL: NCT06618027
Title: Pragmatic Clinic-Based Trial of a Mindfulness Based Intervention for Mood Concerns in Youth With Type 1 Diabetes
Acronym: BREATHE-T1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Barbara Davis Center of Childhood Diabetes, University of Co (Unknown); Colorado State University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000998; 1R01DK137859-01A1 (NIH)
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: type 1 diabetes; adolescents; depression; anxiety
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Intervention, BREATHE-T1D (Experimental): Learning to BREATHE, an existing group-based mindfulness intervention, was adapted in a prior trial, using the input of teens with T1D, to utilize mindfulness as a strategy for supporting the management of T1D. The intervention is 7 sessions, one per week, 60-90 minutes each and teaches mindfulness strategies and promotes connection with other teens with T1D.
  Interventions: Behavioral: BREATHE-T1D
- Diabetes Education and Support, HealthEd-T1D (Placebo Comparator): HealthEd-T1D was designed using input of teens with T1D to be a 6 session, 60 minutes once per week program to promote knowledge and empowerment in diabetes management as well as to encourage connection with other teens with T1D.
  Interventions: Behavioral: HealthEd-T1D

INTERVENTIONS:
Behavioral: BREATHE-T1D — BREATHE-T1D was adapted from Learning to BREATHE, a group mindfulness-based intervention for teens. It teaches mindfulness strategies adapted to be specific and relatable to, teens with T1D to improves symptoms of depression and anxiety as well as diabetes self-management.
  Arms: Mindfulness-Based Intervention, BREATHE-T1D
Behavioral: HealthEd-T1D — HealthEd-T1D is a 6 week, virtual, group based diabetes education group.
  Arms: Diabetes Education and Support, HealthEd-T1D

SUMMARY:
Type 1 diabetes (T1D) is a common chronic illness among children requiring a high degree of self-management for good glycemic control. Adolescents are at risk for poor disease management and health outcomes due to a number of factors, including high rates of depression, anxiety, and stress. Accessing support for these challenges can be a barrier to care, so the current study, BRinging Empowerment and Attention to Teen HEalth-T1D, evaluates the efficacy of a virtual, group-based mindfulness based intervention and a virtual group-based diabetes education intervention on improving symptoms of depression and anxiety, and diabetes self management in teens with T1D. The study also aims to study how these interventions might be implemented in diabetes clinic settings.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is one of the most common chronic illnesses of childhood affecting around 200,000 youth in the US. Youth with T1D are at heightened risk for serious adverse health consequences as compared to their peers without T1D, but treatment adherence markedly reduces this risk. Adolescence is a critical period for determining the course of T1D as treatment adherence and glycemic target achievements deteriorate in adolescence, with ~80% failing to meet glycemic targets. Adolescents' failure to adhere to standards of treatment can result in poor glycemic control (HbA1c >7.0%), which if unaddressed, increases the risk of serious adverse health consequences. Effective intervention to address glycemic control in adolescents with T1D remains elusive. Negative affect-including depression and anxiety-increases during adolescence and is a key contributor to treatment non-adherence and glycemic control above targets. As many as 40% of adolescents with T1D have elevated depression and anxiety symptoms, which likely impact adherence and glycemia through stress-related behavior (e.g., disordered eating, avoidant coping). Trials of effective interventions to decrease negative affect and downstream, stress-related behaviors are critical to improve the health of adolescents with T1D.

Our pilot study adapted a brief group mindfulness-based intervention (MBI) for teens with T1D utilizing stakeholder input and designed with an iterative approach (BREATHE-T1D). Our R34 demonstrated that BREATHE-T1D was highly feasible (100% of eligible teens approached enrolled with a 93% retention rate) and demonstrated outstanding acceptability, with teens participating in 98% of sessions and reporting high value of participation. Those randomized to BREATHE-T1D had evidence of more clinical improvement for depression and HbA1c while those in the health education comparison had stability or worsening of symptoms. Improvements over time were seen in anxiety, diabetes distress, and disordered eating for participants. Existing data from randomized controlled trials (RCT) support the efficacy of MBI for decreasing negative affect and stress-related behavior in adolescents without T1D. The next step is to evaluate the efficacy of BREATHE-T1D in a 2-site study as compared to our health education attention control (HealthEd-T1D). In our R34, providers noted that many adolescents have psychosocial concerns, yet there are grossly inadequate referral sources and a need for integration of efficacious programs into clinic settings. Therefore, it is critical to design interventions for implementation and sustainability and evaluate how the intervention is aligned with infrastructure in real world settings.

The current study is a partnership with Children's National and the University of Colorado to conduct an RCT comparing BREATHE-T1D and HealthEd-T1D in N=200 adolescents 13-17y with >1 year duration of T1D and elevated negative affect. This study is a pragmatic trial to evaluate the efficacy of BREATHE-T1D and methods of implementation of this program into the clinic setting for which it is designed. Given the positive response to the pilot trial, the value of evaluating screening and referral in clinic, increased emphasis on in-clinic screening for mood, anxiety, and disordered eating, and evaluating outcomes relevant to the clinic setting enables both evaluation of efficacy as well as feasibility of clinic implementation. The intervention will be conducted virtually and the trial will employ multi-method assessment of outcomes including self-report, parent-report, and indica-tors of diabetes management (i.e., blood glucose variability via Continuous Glucose Monitors or blood glucose meters and glycemic control via HbA1c). N=200 adolescents will be randomized 1:1 to BREATHE-T1D or HealthEd-T1D and have a baseline assessment, 7 weeks of groups, and follow-ups 3 months and 1 year following baseline.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed for at least 1 year
* Elevated score on depression measure OR elevated score on anxiety measure

Exclusion Criteria:

* Cognitive or developmental delays that restrict ability to complete study interventions or assessments
* Teen not fluent in English
* No other serious medical conditions (e.g., cystic fibrosis, cancer)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-08-06 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | Baseline, 3-, and 12-months post intervention
  Glycemic control will be measured by at home hemoglobin A1c kits as well as downloads of continuous glucose monitor or blood glucose meter data across a 2 week period, with percent of time in range (70-180) calculated and HbA1c used as an indicator of glycemic control over the prior 3 months.
Depression | Baseline, 3-, and 12-months post intervention
  Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D is a self-report scale on symptoms of depression experienced over the prior two weeks. The possible range of scores is 0-60 with higher scores indicating more severe symptoms of depression.

SECONDARY OUTCOMES:
Anxiety | Baseline, 3-, and 12-months post intervention
  Screen for Child Anxiety Related Disorders (SCARED). The SCARED is a self report measure with higher scores indicative of an anxiety disorder.
Disordered Eating | Baseline, 3-, and 12-months post intervention
  Diabetes Eating Problem Survey - Revised (DEPS-R) is a self-report measure that asks about disordered eating behaviors, including those specific to individuals with diabetes. Higher scores indicate more disordered eating symptoms.
Mindfulness | Baseline, 3-, and 12-months post intervention
  Mindful Attention Awareness Scale (MAAS) is a self-report measure assessing how mindful people are in their day to day lives. Higher scores indicate higher levels of dispositional mindfulness.
Mindfulness | Baseline, 3-, and 12- months
  The Five-Factor Mindfulness Questionnaire is a self-report measure that evaluates elements of mindfulness, including the following aspects: observing, describing, acting with awareness, nonreactivity, and non-judgement. Higher scores indicate a higher level of mindfulness.
Stress | Baseline, 3-, and 12-months post intervention
  PROMIS Stress Scale is a brief self-report measure that asks about experiences of stress over the past 2 weeks. Higher scores indicate more experiences of stress.
Executive Functioning | Baseline, 3-, and 12-months post intervention
  Parent report Behavior Rating Inventory of Executive Function (BRIEF). The BRIEF uses parent report of adolescent executive function, or the ability to plan, organize, and other aspects of executive function. Higher scores indicate the presence of executive functioning challenges.
Negative Urgency | Baseline, 3-, and 12-months post intervention
  UPPS-P Negative Urgency scale is a self-report scale which assesses impulsive behavior, particularly when experiencing negative mood. Higher scores indicate greater challenge with acting impulsively when upset.
Avoidant Coping | Baseline, 3-, and 12-months post intervention
  Responses to Stress Questionnaire - Diabetes (RSQ-D). The Responses to Stress Questionnaire is a self- and parent- reported measure assessing presence of stressors, some of which are specific to having diabetes, and what coping strategies are used to manage these. Higher scores indicate more use of various coping strategies.
Diabetes Distress | Baseline, 3-, and 12-months post intervention
  Problem Areas in Diabetes Scale - Teen (PAID-T). The PAID-T is a self-report measure that assesses a teen's perspective on how much distress they experience as a result of having or managing type 1 diabetes. HIgher scores indicate greater levels of diabetes-related distress.
Diabetes Self-Management | Baseline, 3-, and 12-months post intervention
  Self Care Inventory (SCI). The SCI is a self-report measure on how much the teen adheres to medical recommendations to self-manage their diabetes. Higher scores indicate the presence of more self-management behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Mackey, PhD, Principal Investigator — children's national hospital
Locations (2):
- United States (2):
  - Barbara Davis Center, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No